CLINICAL TRIAL: NCT07183241
Title: Comparación Entre Ingreso Hospitalario y Hospitalización Domiciliaria y Análisis de Una Intervención Multicomponente en Adultos Mayores: Ensayo Clínico Aleatorizado
Brief Title: Hospital-to-Home Rehabilitation Through Exercise and Cognitive Training
Acronym: H-REACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pública de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI_2025/34
Record Dates: First submitted 2025-06-10; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-06

CONDITIONS: Acute Hospitalization
Keywords: acute hospitalization; older adults; exercise; hospital at home; cognitive
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This research project is structured in two phases: an initial observational phase comparing hospital admission and hospital at home, and a subsequent randomized controlled trial phase assessing the efficacy of a multicomponent post-hospitalization intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent intervention (Experimental): Physical exercise and cognitive exercises
  Interventions: Behavioral: Physical exercise and cognitive exercises
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Physical exercise and cognitive exercises — The intervention will be based on the Vivifrail program, which is a multicomponent physical exercise program designed specifically for older adults.
  Arms: Multicomponent intervention

SUMMARY:
This research project is structured in two phases: an initial observational phase and a subsequent randomized controlled trial (RCT) phase. The goal of the observational phase is to compare hospital admission and Hospital at Home (HaH). The objective of the RCT is to assess the effectiveness of a multicomponent intervention following acute hospitalization in older adults. The main questions it aims to answer are:

* What are the differences between hospital admission and HaH in sedentary and physical activity levels?
* What are the effects of a multicomponent intervention following acute hospitalization in older adults?

Researchers will compare a post-discharge multicomponent intervention to usual care to see the effects on physical and cognitive function.

Participants will receive a home-based cognitive and physical exercise intervention or usual care.

ELIGIBILITY:
Inclusion Criteria:

* Older adults admitted to the hospital or Hospital at Home (HaH) due to an acute illness.
* Residents of Navarre.
* Willingness to participate on a voluntary basis.
* Ability to ambulate with or without assistance.
* Ability to communicate and collaborate with the research staff.

Exclusion Criteria:

* Acute illness that does not allow the assessment and practice of physical exercise during the study.
* Medical contraindication for the practice of physical exercise.
* Severe dementia.
* Refusal to sign the informed consent form by the patient, accompanying person, or legal guardian.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Physical function | Within the first 24-48 hours of acute care admission (in hospital or home hospitalization), pre-intervention baseline, and immediately after the intervention.
  Short Physical Performance Battery (SPPB): scores range from 0 to 12, with higher scores indicating better physicalfunction.
Cognitive function | Within the first 24-48 hours of acute care admission (in hospital or home hospitalization), pre-intervention baseline, and immediately after the intervention.
  Mini-Mental State Examination (MMSE): scores range from 0 to 30, with higher scores indicating better cognitive function.
Physical activity | During hospital stay or during home-base hospitalization .
  Physical activity will be assessed with a Firstbeat device (format: hh:mm:ss).
Sedentarism | During hospital stay or during home-based hospitalization.
  Sedentarism will be assessed with a Firstbeat device (format: hh:mm:ss).

SECONDARY OUTCOMES:
Health-related quality of life (HRQOL) | Pre-intervention baseline and immediately after the intervention.
  EQ-5D-5L provides a health profile that is converted to a utility index, in which 0 is equivalent to death and 1 indicates perfect health. Additionally, the EQ-VAS ranges from 0 to 100, with higher scores indicating better health.
Heart rate variability | During hospital stay or during home-based hospitalization.
  Heart rate variability will be assessed usign a Firstbeat device.
Handgrip strength | Within the first 24-48 hours of acute care admission (in hospital or home hospitalization), pre-intervention baseline, and immediately after the intervention.
  Handgrip strength will be measured using a handgrip dynamometer.
Sleep quantity | During hospital stay or during home-based hospitalization.
  Sleep duration will be recorded (format: hh:mm:ss).
Sleep quality | During hospital stay or during home-based hospitalization.
  The heart rate variability parameter RMSSD (measured in ms) will be assessed during sleep.
Energy expenditure | Within the first 24-48 hours of acute care admission (in hospital or home hospitalization), pre-intervention baseline, and immediately after the intervention.
  Energy expenditure (kcal) will be assessed in with a Firstbeat device.
Rate of hospital readmissions | 3 months, 6 months, and 12 months post-discharge.
  Number of readmissions of each patient will be registered using the information from the medical records.
Rate of falls | 3 months, 6 months, and 12 months post-discharge.
  The number of falls for each patient will be recorded through follow-up phone calls.
Incidence of mortality | 3 months, 6 months, and 12 months post-discharge.
  Number of deaths will be registered using the information from the medical records.
Rate of emergency visits | 3 moths, 6 months, and 12 months post-discharge.
  Number of emergency visits will be registered using the information from the medical records.
Prescribed pharmacologic treatment | Within the first 24-48 hours of acute care admission (in hospital or home hospitalization), pre-intervention baseline, and immediately after the intervention.
  All medications prescribed to each patient will be recorded using the information from the medical records.
Cost-effectiveness | At pre-intervention baseline, at 3 months post-discharge, at 6 months post-discharge, and at 12 months post-discharge.
  Cost-effectiveness will be assessed by calculating the cost per Quality-Adjusted Life Year (QALY) gained.

IPD SHARING:
Plan to Share IPD: Undecided